CLINICAL TRIAL: NCT04244799
Title: Evaluating the Impact of Behavioral Nudges on Student Independent Hand-washing Practices in Elementary Schools in the Philippines
Brief Title: Evaluating the Impact of Behavioral Nudges on Student Hand-washing in Elementary Schools in the Philippines
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IDinsight (Other)
Collaborators: United States Agency for International Development (USAID) (U.S. Federal Agency); UNICEF (Other); Philippines Department of Education (Unknown)
Responsible Party: Principal Investigator, Haijing Huang, Economist, IDinsight
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 005
Record Dates: First submitted 2020-01-21; First posted 2020-01-28 (Actual); Last update posted 2020-03-27 (Actual); Status verified 2020-03

CONDITIONS: Hand Disinfection
Keywords: Handwashing; Behavioral nudge; Contextual cue; Philippines; Health behavior; Nudge; Environmental cue; Behavior change
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Behavioral nudges (Experimental): Schools randomized to this arm will receive the behavioral nudges intervention and the Philippines Department of Education national WASH in Schools (WinS) policy.
  Interventions: Behavioral: Behavioral nudges; Behavioral: National WASH policy
- Control group (Active Comparator): Schools in the control group will not receive handwashing nudges but will receive DepEd's national WASH in Schools (WinS) policy.
  Interventions: Behavioral: National WASH policy

INTERVENTIONS:
Behavioral: Behavioral nudges — Behavioral nudges include the following:
  1. Colorful pathway overlaid with footprints leading from the toilet to the handwashing station
  2. Rotating posters in toilet areas with messages targeting behavioral motivators for handwashing (disgust, social affiliation)
  3. Sticker of a pair of eyes placed above the handwashing station
  4. Soap dish with an arrow beside it on the sink or counter to remind children to wash their hands with soap
  Arms: Behavioral nudges
Behavioral: National WASH policy — The Philippines' Department of Education National WASH in Schools (WinS) policy promotes "correct hygiene and sanitation practices among school children and a clean environment in and around schools" and includes initiatives related to infrastructure, knowledge, and behavior change, but does not include other programs with an explicit focus on handwashing promotion.

SUMMARY:
This study evaluates the impact of school-based behavioral "nudges" installed in toilets and handwashing facilities on handwashing behavior among students in the Philippines. Nudges include: visible signage crafted to trigger behavioral motivators for handwashing; colorful pathway overlaid with footprints leading from the toilet to the handwashing station; sticker of a pair of eyes placed above the handwashing station; soap dish with an arrow beside it on the sink or counter to remind children to wash their hands with soap. The study's main hypothesis is that behavioral nudges will increase the percentage of students who wash their hands with water and soap after toilet use by 7 percentage points or more among schools where nudges were installed compared to control schools without nudges. The study is taking place in public primary schools in Zamboanga Del Norte, Philippines between October 2019 and May 2020.

DETAILED DESCRIPTION:
The impact of the behavioral nudge intervention will be evaluated using a cluster randomized controlled trial (RCT). The investigators will randomly select 132 Department of Education (DepEd) schools across Zamboanga Del Norte province to comprise the study sample. 66 schools will be assigned to the treatment group, and 66 schools to the control group. Treatment schools will receive the behavioral nudge intervention, while control group will not. Both treatment and control schools will receive DepEd's national WASH in Schools (WinS) policy. WinS promotes "correct hygiene and sanitation practices among school children and a clean environment in and around schools" and includes initiatives related to infrastructure, knowledge, and behavior change, but does not include other programs with an explicit focus on handwashing promotion.

Four months after installing nudges, enumerators will conduct structured observations in study schools, observing whether pupils wash their hands with soap, wash without soap, or do not wash, after they have used classroom toilets. This will be used to estimate the causal impact of the nudges intervention on rates of independent handwashing with water and soap after toilet use.

ELIGIBILITY:
Inclusion criteria:

* Water for handwashing is available at the school for at least certain days of the week
* The overall pupil to toilet ratio equals 100 or lower
* School has at least one individual handwashing station or group handwashing station
* School is situated in a district deemed safe by DepEd
* School does not have any planned WASH programming in the upcoming 2019-20 school year beyond standard WinS activities

Exclusion Criteria:

* Water for handwashing is not available at the school for all days of the week
* The overall pupil to toilet ratio equals over 100
* School does not have either an individual handwashing station nor a group handwashing station
* School is situated in a district deemed unsafe by DepEd
* School has at least one planned WASH programming in the upcoming 2019-20 school year beyond standard WinS activities

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 99 (Actual)
Dates: Start 2020-02-10 (Actual); Primary Completion 2020-03-02 (Actual); Study Completion 2020-03-02 (Actual)

PRIMARY OUTCOMES:
The probability that a student was observed to wash their hands with soap and water after toilet use | 4 months
  Unit of analysis: student
The probability that a student was observed to wash their hands with water after toilet use | 4 months
  Unit of analysis: student

SECONDARY OUTCOMES:
The number of functioning handwashing facilities at the school | 4 months
  Unit of analysis: school
The number of functioning handwashing facilities with soap and water at the school | 4 months
  Unit of analysis: school
The probability that a toilet facility has a nearby functioning handwashing facility | 4 months
  Unit of analysis: toilet facility. A "nearby" handwashing facility means inside the classroom for toilet facilities located inside classrooms and within 10 meters of toilet facilities located outside classrooms.
The probability that a toilet facility has a nearby functioning handwashing facility with water and soap | 4 months
  Unit of analysis: toilet facility. A "nearby" handwashing facility means inside the classroom for toilet facilities located inside classrooms and within 10 meters of toilet facilities located outside classrooms.

CONTACTS AND LOCATIONS:
Overall Officials: Haijing Huang, PHD, Principal Investigator — IDinsight; Meghan Battle, MPH, Principal Investigator — IDinsight
Locations (1):
- IDinsight, Manila, Philippines

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Statistical Analysis Plan (2020-01-20): https://cdn.clinicaltrials.gov/large-docs/99/NCT04244799/SAP_000.pdf